CLINICAL TRIAL: NCT00036946
Title: An Open-Label, Sequential Cohort Dose-Escalation Safety, Tolerability And Pharmacokinetic Study Of VEGF Trap In Patients With Incurable, Relapsed Or Refractory Solid Tumors Or Lymphoma
Brief Title: VEGF Trap in Treating Patients With Relapsed or Refractory Solid Tumors or Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: REGENERON-VGFT-ST-0103; MSKCC-01131; CDR0000069343 (Registry Identifier: PDQ (Physician Data Query)); NCI-G02-2065
Record Dates: First submitted 2002-05-13; First posted 2003-01-27 (Estimated); Last update posted 2016-06-03 (Estimated); Status verified 2016-06

CONDITIONS: Lymphoma; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; stage IV adult diffuse small cleaved cell lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult immunoblastic large cell lymphoma; stage IV adult lymphoblastic lymphoma; stage IV adult Burkitt lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent adult Burkitt lymphoma; stage IV mantle cell lymphoma; recurrent mantle cell lymphoma; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; stage IV small lymphocytic lymphoma; stage IV marginal zone lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Follicular; Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Burkitt Lymphoma; Lymphoma, Mantle-Cell; Lymphoma, B-Cell, Marginal Zone; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — aflibercept

INTERVENTIONS:
Biological: ziv-aflibercept

SUMMARY:
RATIONALE: VEGF Trap may stop the growth of solid tumors or non-Hodgkin's lymphoma by stopping blood flow to the cancer.

PURPOSE: Phase I trial to study the effectiveness of VEGF Trap in patients who have relapsed or refractory solid tumors or non-Hodgkin's lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the safety and tolerability of VEGF Trap in patients with incurable relapsed or refractory solid tumors or non-Hodgkin's lymphoma.
* Determine the maximum tolerated dose of this drug in these patients.
* Determine the pharmacokinetics of this drug in these patients.
* Evaluate the ability of this drug to bind and inactivate circulating vascular endothelial growth factor (VEGF) in these patients.
* Determine the dosing regimen that is optimal for neutralization of circulating VEGF in these patients.
* Determine whether antibodies to this drug develop in these patients.
* Assess, preliminarily, the ability of this drug to alter tumor vascular permeability and tumor growth in these patients.

OUTLINE: This is a dose-escalation study.

Patients receive VEGF Trap subcutaneously once daily on days 1, 29, 36, 43, 50, 57, and 64 in the absence of disease progression or unacceptable toxicity.

Cohorts of 1-6 patients receive escalating doses of VEGF Trap until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose-limiting toxicity. Once the MTD is determined, 5 additional patients are treated at the MTD.

Patients are followed at 1 and 4 weeks.

PROJECTED ACCRUAL: A maximum of 30 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed incurable primary or metastatic solid tumor or non-Hodgkin's lymphoma

  * Relapsed after or is refractory (e.g., unresectable) to at least 2 standard chemotherapy regimens and rituximab
  * No standard curative surgery, chemotherapy, immunotherapy, other antitumor therapy, or radiotherapy options exist
* No known or suspected squamous cell carcinoma of the lung
* No prior or concurrent CNS (brain or leptomeningeal) metastases
* No prior or concurrent primary intracranial tumor by MRI or CT scan

PATIENT CHARACTERISTICS:

Age:

* 25 and over

Performance status:

* ECOG 0-2

Life expectancy:

* Not specified

Hematopoietic:

* WBC at least 3,500/mm^3
* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* Hemoglobin at least 9.0 g/dL
* No other severe or uncontrolled hematologic condition

Hepatic:

* Bilirubin no greater than 1.5 times upper limit of normal (ULN)
* AST and ALT no greater than 2 times ULN
* Alkaline phosphatase no greater than 2 times ULN
* PT, PTT, and INR normal

Renal:

* Creatinine no greater than ULN
* No 1+ or greater proteinuria
* No other severe or uncontrolled renal condition

Cardiovascular:

* Electrocardiogram normal
* LVEF normal by echocardiogram or MUGA scan within the past 12 months or since completion of prior anthracycline
* No severe or uncontrolled cardiovascular condition
* No New York Heart Association class III or IV heart disease
* No active coronary artery disease, angina, congestive heart failure, or arrhythmia
* No myocardial infarction within the past 6 months
* No prior or concurrent peripheral vascular disease, including:

  * Angiographically or ultrasonographically documented arterial or venous occlusive event
  * Symptomatic claudication
* No untreated or uncontrolled hypertension
* No treated blood pressure more than 160/100 mm Hg on at least 3 repeated determinations on separate days within the past 6 weeks
* No symptomatic orthostatic hypotension

Pulmonary:

* No severe or uncontrolled pulmonary condition
* No pulmonary embolism

Other:

* No prior hypersensitivity reactions to any recombinant proteins (e.g., VEGF Trap)
* No severe or uncontrolled gastrointestinal, immunological, or musculoskeletal condition
* No severe or uncontrolled psychiatric or adverse social circumstance that would preclude study
* No active infection requiring antibiotics
* HIV negative
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective double-barrier contraception during and for at least 3 months after study

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* See Disease Characteristics
* At least 3 weeks since prior immunotherapy
* No concurrent epoetin alfa, filgrastim (G-CSF), or sargramostim (GM-CSF)

Chemotherapy:

* See Disease Characteristics
* At least 3 weeks since prior chemotherapy

Endocrine therapy:

* No concurrent adrenal corticosteroids, except low doses as replacement therapy in patients who have previously received suppressive doses or for adrenal insufficiency
* No concurrent systemic hormonal contraceptive agents

Radiotherapy:

* See Disease Characteristics
* At least 3 weeks since prior radiotherapy

Surgery:

* See Disease Characteristics
* At least 3 weeks since prior surgery (except fine needle biopsy/aspiration or removal/biopsy of a skin lesion)
* No prior surgical procedure for correction or prophylaxis of peripheral vascular insufficiency or cerebral ischemic events

Other:

* Recovered from prior therapy
* At least 6 months since prior treatment for acute congestive heart failure
* At least 30 days since prior investigational drugs
* No concurrent standard or other investigational anticancer agents
* No concurrent herbal supplements ("nutraceuticals")
* No concurrent anticoagulant or antiplatelet drugs, (e.g., warfarin, heparin, aspirin, or other non-steroidal anti-inflammatory drugs) except selective cyclo-oxygenase-2 (COX-2) inhibitors for analgesia
* No concurrent COX-2 inhibitors for tumor treatment or prophylaxis

Ages: 25 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2001-11; Primary Completion 2002-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jakob Dupont, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

REFERENCES:
- [Result] Dupont J, Schwartz L, Koutcher J, et al.: Phase I and pharmacokinetic study of VEGF Trap administered subcutaneously (sc) to patients (pts) with advanced solid malignancies. [Abstract] J Clin Oncol 22 (Suppl 14): A-3009, 197s, 2004.
- [Result] Dupont J, Camastra D, Gordon MS, et al.: Phase 1 study of VEGF Trap in patients with solid tumors and lymphoma. [Abstract] Proceedings of the American Society of Clinical Oncology 22: A-776, 2003.
- [Result] Tew WP, Gordon M, Murren J, Dupont J, Pezzulli S, Aghajanian C, Sabbatini P, Mendelson D, Schwartz L, Gettinger S, Psyrri A, Cedarbaum JM, Spriggs DR. Phase 1 study of aflibercept administered subcutaneously to patients with advanced solid tumors. Clin Cancer Res. 2010 Jan 1;16(1):358-66. doi: 10.1158/1078-0432.CCR-09-2103. Epub 2009 Dec 22. PMID 20028764